CLINICAL TRIAL: NCT01188317
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Effect of Ibuprofen on Top of Multiple Doses of 150 µg Aleglitazar Once Daily on Renal Function, Renin-angiotensin System, and Pharmacokinetics of Both Compounds in Healthy Subjects
Brief Title: A Study of Aleglitazar in Combination With Ibuprofen in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25330
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: aleglitazar; Drug: ibuprofen
- 2 (Placebo Comparator)
  Interventions: Drug: placebo; Drug: ibuprofen

INTERVENTIONS:
Drug: aleglitazar — repeated daily doses
  Arms: 1
Drug: placebo — repeated daily doses
  Arms: 2
Drug: ibuprofen — repeated daily doses

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group study will investigate the safety and tolerability, and the effect of aleglitazar in combination with ibuprofen on renal function, renin-angiotensin system and pharmacokinetics in healthy volunteers. Volunteers will be randomized to receive daily doses of aleglitazar or placebo in combination with ibuprofen. The anticipated time on study drug is 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged 40 to 65 years inclusive
* Body Mass Index (BMI) between 18 and 35 kg/m2 inclusive
* Females of child-bearing potential must be willing to use two acceptable methods of contraception during the study and at least 3 months before start of the study
* Non-smoker or currently smoking less than 5 cigarettes (or equivalent amount of other tobacco products) per day and is willing and able to stop smoking during the period in study center
* Volunteer drinks no more than 3 cups of coffee, tea or soft drinks per day and is willing and able to stop drinking coffee, tea and soft drinks during the period in study center

Exclusion Criteria:

* Any clinically relevant abnormal laboratory test results at screening
* Volunteer has taken any prescribed, herbal or over-the-counter medication within 2 weeks prior to first dosing
* A history of any clinical significant gastro-intestinal, cardiovascular, musculoskeletal, endocrine, hematological, psychiatric, renal, hepatic, bronchopulmonary or neurological conditions or lipid disorders
* A positive test for human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B or hepatitis C
* History of intolerance to non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin, history of gastric or duodenal ulceration, personal or family history of abnormal clotting or bleeding

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To assess the effect of ibuprofen in combination with aleglitazar on measured glomerular filtration rate | 12 weeks

SECONDARY OUTCOMES:
To investigate the effect of ibuprofen in combination with aleglitazar on renal plasma flow, filtration fraction and estimated glomerular filtration rate | 12 weeks
To investigate the effect of ibuprofen in combination with aleglitazar on renin-angiotensin system and on anti-diuretic hormone | 12 weeks
To investigate the pharmacokinetics of aleglitazar and ibuprofen when co-administered | 12 weeks
To investigate safety and tolerability of aleglitazar | 12 weeks
To investigate the effect of aleglitazar in combination with ibuprofen on electrolytes and osmolality clearances | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Omaha, Nebraska, United States